CLINICAL TRIAL: NCT04758052
Title: Bedside Gastrostomy With Simultaneous Tracheostomy Effect On Outcomes Of Neurocritically-Ill Patients (Proof Of Concept Study)
Brief Title: Tracheostomy With Bedside Simultaneous Gastrostomy Vs Usual Care Tracheostomy And Delayed Gastrostomy Placement
Acronym: BEGASTON
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator change in institution
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020V0278
Record Dates: First submitted 2021-02-04; First posted 2021-02-17 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Acute; TBI; Neuromuscular Diseases; Status Epilepticus; Coma; Cerebrovascular Disorders; Spinal Cord Injuries; Neurological Injury; Neurologic Injury
MeSH Terms: conditions — Stroke; Neuromuscular Diseases; Status Epilepticus; Coma; Cerebrovascular Disorders; Spinal Cord Injuries; Trauma, Nervous System

STUDY DESIGN:
Intervention Model Description: single-center prospective randomized open-label blinded endpoint proof-of-concept study to assess the effect of TSG versus usual care TDG placement on outcomes among neurocritically-ill patients.
Masking Description: blinded endpoint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simultaneous tracheostomy with gastrostomy (TSG) (Experimental): This arm include the patients assigned to placement of gastrostomy immediately after tracheostomy.
  Interventions: Other: Timing of placement
- non-simultaneous or delayed approach tracheostomy and gastrostomy (TDG) (No Intervention): This arm include the patients who proceed with "usual care" placement of tracheostomy and gastrostomy as per Neurocritical care Unit service standard.

INTERVENTIONS:
Other: Timing of placement — Simultaneous placement of tracheostomy and gastrostomy
  Arms: simultaneous tracheostomy with gastrostomy (TSG)

SUMMARY:
There is currently no prospective study analyzing the effect of tracheostomy with bedside simultaneous gastrostomy versus tracheostomy with delayed gastrostomy placement (TSG versus TDG) on the outcomes of neurocritically-ill patients. The investigators will study TSG via concomitant PDT and PUG procedures, while TDG will occur per usual care. This study is a prospective randomized open-label blinded endpoint study to assess the effect of tracheostomy with bedside simultaneous gastrostomy (TSG) versus the usual care of tracheostomy with delayed gastrostomy (TDG) placement on outcomes of neurocritically-ill patients.

DETAILED DESCRIPTION:
The practice of performing tracheostomy and gastrostomy simultaneously has been reported since the 1980s. The safety and feasibility of simultaneous tracheostomy with gastrostomy (TSG), compared to non-simultaneous or delayed approach (TDG), among neurocritically-ill patients have been reported by various case series and retrospective cohort studies.The timing of tracheostomy generally among neurocritically-ill patients varies from early <5 days or late >7 -10 days. There are currently no guidelines specifically on neurocritically-ill patients and the timing of gastrostomy placement however, it is generally recommended to wait 2-3 weeks as a time limited trial however, there are patients that are able to leave the hospital with the main limitation as being the feeding access. Although it has been suggested to consider tracheostomy to become an indication for gastrostomy this has not been widely accepted although there is an increase in awareness of the TSG approach especially in patients with neurologic conditions.

Tracheostomy have been traditionally indicated include airway obstruction associated with infection, malignancy, injury, sleep apnea and vocal cord dysfunction, prolonged intubation, facilitate weaning from mechanical ventilation, pulmonary hygiene and aspiration.

Gastrostomy tubes have been considered as standard of care for patients requiring alternate forms of long-term enteral feeding. Other indications include long-term nutrition support associated with neurologic or spinal cord deficits, primary swallowing dysfunction, facial or pharyngeal injuries, malignancy of the head and neck and the esophagus, gastric decompression. Approaches available to perform tracheostomy include open, percutaneous tracheostomy, percutaneous dilatational tracheostomy (PDT); Percutaneous Radiologic Tracheostomy and percutaneous ultrasound tracheostomy. Gastrostomy is a temporary or permanent controlled fistula from the lumen of the stomach to the skin. For gastrostomy, approaches include open surgical gastrostomy (SG) or Stamm gastrostomy, Percutaneous endoscopic gastrostomy (PEG), Percutaneous Radiologic gastrostomy (PRG) and Percutaneous Ultrasound gastrostomy (PUG).

In a retrospective cohort study on the outcomes of neurocritically-ill patients who have undergone TSG versus delayed gastrostomy TDG (non-simultaneous tracheostomy and gastrostomy), the patients undergoing TSG had shorter Neurocritical Care Unit (NCCU) length of stay (LOS), hospital LOS, overall hospital cost and higher pre-discharge prealbumin levels. In another study examining the effect of early gastrostomy tube placement on stroke patients, it was found that early gastrostomy tube placement was associated with shorter LOS and higher odds of home or acute rehabilitation discharge disposition. In a retrospective study on intracerebral hemorrhage and subarachnoid hemorrhage patients, it was found that tracheostomy was associated with ICU LOS with almost a 10-day difference if tracheostomy is placed before 7 days or after 14 days. They also found a 6- day difference in overall length of stay between those who had the gastrostomy tubes placed before 7 days or after 14 days. Importantly they saw that the timing of tracheostomy and gastrostomy placement was not associated with mortality. In practice, usual care favors delayed gastrostomy due to availability of imaging resources, proceduralist coordination, and provider preference. Bedside PEG requires the availability of specialized mobile endoscopic equipment and physicians trained in upper endoscopy. In a retrospective study of TSG, among the most common reason for procedural delays were coordination with GI service for performance of PEG. Further, mobile endoscopes are expensive and uncommon across the healthcare system, thus preventing PEG from practical generalizability as an early gastrostomy technique. TSG has been performed using standard PDT and PUG. Because PUG utilizes point-of-care ultrasound (POCUS) technology readily available at the bedside it is a generalizable method for early gastrostomy. Finally, direct comparative evidence to support guidelines for TSG over TDG do not exist. In the absence of clear guidelines, provider preference permits delayed gastrostomy decisions.There is currently no prospective study analyzing the effect of tracheostomy with bedside simultaneous gastrostomy versus tracheostomy with delayed gastrostomy placement (TSG versus TDG) on the outcomes of neurocritically-ill patients. To analyze the effect on patient outcomes of early intervention (TSG versus TDG), a pragmatic randomized clinical trial is needed. The investigators will study TSG via concomitant PDT and PUG procedures, while TDG will occur per usual care. This study is a prospective randomized open-label blinded endpoint study to assess the effect of tracheostomy with bedside simultaneous gastrostomy (TSG) versus the usual care of tracheostomy with delayed gastrostomy (TDG) placement on outcomes of neurocritically-ill patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old- 85 years old
* Admitted under the NSICU service
* Shared-decision making with surrogate decision maker and primary neuro-intensivist agreement to proceed with tracheostomy and gastrostomy with documented discussion.
* have indications for tracheostomy and gastrostomy
* Subjects or their SDM or legally authorized representative (LARs) must voluntarily provide informed consent prior to the initiation of any study-specific procedure in a form approved by an independent IRB. In the absence of subject's ability to provide informed consent, informed consent must be given by a person who has the legal right to act on behalf of the subject in accordance with local laws.

Exclusion Criteria:

* Patients who require tracheostomy only or gastrostomy only
* history of prior gastrostomy, tracheostomy, laryngectomy, gastrostomy prior to tracheostomy decision, known head and neck and gastrointestinal abnormality (cancer, congenital abnormality, anatomic variants)
* withdrawal of care, a transfer from another service or hospital if patient has been there for >24hr.
* known social discharge issues anticipating hospital stay >100 days
* Patients with nonsurvivable injuries, anticipated mortality <72 hours
* standard of care contraindications for either bedside tracheostomy and gastrostomy
* Absolute contraindications for gastrostomy: gastric outlet obstruction, significant gastroparesis, significant gastroesophageal reflux, a proximal high-output entercutaneous fistula
* Standard Contraindications for percutaneous gastrostomy technique: ascites, morbid obesity and esophageal and gastric pathology
* Standard Contraindications for either PEG or PUG procedures
* Standard Contraindications to percutaneous dilational tracheostomy: Gross anatomical distortion of the neck, previous neck surgery , burns, radiotherapy, unstable or rigid cervical spine, tracheal distortion, stenosis, or malacia, morbid obesity (BMI >35kg/m2), massive thyroid gland or vessels in the operation field on ultrasound, hemodynamic instability, refractory intracranial hypertension, hemodynamic instability, Coagulopathy (Aptt>50s, INR>1.5, platelet count <50,000μL, emergency need for a tracheostomy or need for a permanent tracheostoma, very difficult airway management
* Pregnancy
* Life expectancy less than three-weeks
* Goals of care disagreement between care team and LAR
* braindead
* LAR preferred procedures placed in LTAC

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
ICU length of stay | during hospital stay, assessed up to 10 days
  total number of midnights a patient is in the ICU for the duration of their hospital stay

SECONDARY OUTCOMES:
hospital length of stay | during hospital stay, assessed up to 10 days
  total number of midnights a patients is in the hospital for the encounter that the patient
nutritional metrics | up to 14 days before the procedure and up to 14-days before discharge
  pre-albumin, albumin, caloric requirements met
procedural analgo-sedation used | intraprocedure
  total dosage of analgo-sedation used
all-cause mortality | during hospital stay, assessed up to 10 days
  proportion of patients who expired due to all-causes
swallow function return | during hospital stay, assessed up to 10 days
  presence, and time to minimal nectar thickened diet is allowed
discharge disposition | during hospital stay, assessed up to 10 days
  discharge location (acute rehabilitation, home, LTAC, nursing home, transferred, expired)
Functional outcome | at discharge, assessed up to 6-months
  Glasgow Outcome Scale Extended, Minimum score =1, Maximum score= 8, lower score is worse
total analgo-sedation dose and duration in the ICU | within ICU-stay, assessed up to 10 days
  total analgo-sedation dosages (infusion and boluses)
proportion of ventilator acquired pneumonia before and after procedures | within ICU stay, assessed up to 10-days
  according to updated CDC definition (https://www.cdc.gov/nhsn/PDFs/pscManual/6pscVAPcurrent.pdf)
overall ICU and hospital cost | within in-hospital stay, assessed up to 10-days
  total ICU cost estimated by LOS and severity-derived-diagnosis-related groups [DRG] multiplicator of each patient (Bösel et al., 2013) and total hospital cost at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Christa O'Hana S. Nobleza, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Undecided